CLINICAL TRIAL: NCT05528341
Title: Clinical Investigation of NKG2D-CAR-NK92 Chimeric Antigen Receptor Modified NK92 Cells in the Treatment of Relapsed/Refractory Solid Tumors
Brief Title: NKG2D-CAR-NK92 Cells Immunotherapy for Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Henan Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNK-102
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Relapsed/Refractory Solid Tumors
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NKG2D-CAR-NK92 cells immunotherapy (Experimental): Preparation of NKG2D-CAR-NK92 cells suspended in saline solution.
  Interventions: Biological: NKG2D-CAR-NK92 cells

INTERVENTIONS:
Biological: NKG2D-CAR-NK92 cells — NKG2D-CAR-NK92 cells will be administered intravenously over 1h. The starting dose of NKG2D-CAR-NK92 cells will be 0.5×10^6-2×10^6/kg, twice a week. The first evaluation of the efficacy after 3 weeks of treatment.

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and effects of NKG2D-CAR-NK92 infusions in the treatment of relapsed/refractory solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 75 years old, male or female.
2. Histopathology confirmed the diagnosis of malignant tumors (including breast cancer, lung cancer, gastric cancer, ovarian cancer, cervical cancer, renal carcinoma, malignant melanoma, osteosarcoma and lymphoma).
3. Expected survival time ≥3 months.
4. Disease must be measurable according to the corresponding guidelines.
5. Fail or unwilling to receive third-line treatment.
6. ECOG: 0-2.
7. The last cytotoxic drug, radiotherapy or surgery≧4 weeks.
8. HB≧90g/L, ANC≧1.5×10^9/L, PLT≧80×10^9/L, TBIL≦1.5×upper limit of normal, ALT/AST≦2.5×upper limit of normal, ALT/AST≦5×upper limit of normal if have liver metastasis, Cr≦1.5×upper limit of normal or CCr≧60ml/min.
9. Women of childbearing age must be tested negative for pregnancy within 7 days, and subjects of childbearing age must use appropriate contraception during both the trial and for 3 months after the test;
10. Written informed consent form must be signed before enrollment.
11. Patient with MICA/B+ cell tumors confirmed by pathology and histology.

Exclusion Criteria:

1. The patient has other malignancies or has been diagnosed with other malignancies within the last 5 years (except clinically cured carcinoma in situ of the cervix, basal cell or squamous cell skin cancer, and thyroid papillary carcinoma).
2. Patients with brain metastases with symptoms or with symptom control for less than 3 months.
3. Active autoimmune disease.
4. Severe autoimmune diseases or congenital immunodeficiency.
5. Concomitant serious infection or other serious underlying medical condition.
6. Active hepatitis patients (including hepatitis B and C).
7. History of severe immediate hypersensitivity to any of the biological products including penicillin.
8. Drug abuse, medical, psychological or social conditions that may interfere with a subject's participation in the study or evaluation of the results of the study.
9. Simultaneous participation in another clinical trial within 4 weeks.
10. Cell therapy or gene therapy in the previous 1 month.
11. A history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency disease, or a history of organ transplantation.
12. Investigator considers that the subject has any clinical or laboratory abnormalities or compliance problems and is not suitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events evaluated with CTCAE, version 4.0 | 3 months
  Safety evaluation
Objective Response Rate | up to one year
  Solid tumors to NKG2D-CAR-NK92 cells infusions

SECONDARY OUTCOMES:
Disease Control Rate | up to one year
Progression-free Survival | up to one year
Overall Survival | up to one year
Quality of Life Score | up to one year
  We use the 26 items self-rating questionnaire WHOQOL-BREF to assess the Quality of Life Score, which measures physical health, psychological health, social relationships, and environment during the last two weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- The first Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan, China

IPD SHARING:
Plan to Share IPD: No